CLINICAL TRIAL: NCT03218579
Title: Endoscopic Assessment and Prediction of Microbiome-modifying Interventions
Acronym: microbiome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-12-ZH-658-CTIL
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Gut Microbiome; Antibiotic Side Effect
Keywords: microbiome; intestinal bacteria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervention (No Intervention): No intervention after antibiotic treatment.
- Probiotic microbiome rehabilitation (Active Comparator): Probiotic treatment after antibiotic treatment.
  Interventions: Dietary Supplement: Probiotic treatment
- Bacteriotherapy microbiome rehabilitation (Active Comparator): Bacteriotherapy after antibiotic treatment.
  Interventions: Biological: Bacteriotherapy

INTERVENTIONS:
Dietary Supplement: Probiotic treatment — 4 weeks of probiotic treatment after 7 days of antibiotics (Metronidazole+Ciprofloxacin)
  Arms: Probiotic microbiome rehabilitation
Biological: Bacteriotherapy — Bacteriotherapy (autologous fecal microbiota transplantation) after 7 days of antibiotics (Metronidazole+Ciprofloxacin)
  Arms: Bacteriotherapy microbiome rehabilitation

SUMMARY:
The investigators would like to examine the extent of gut microbiome rehabilitation in healthy people after the consumption of antibiotics.

Outcomes of probiotic treatment versus bacteriotherapy will be compared.

DETAILED DESCRIPTION:
The investigators would like to examine the extent of rehabilitation of the composition and functioning of the intestinal bacteria in healthy people after the consumption of antibiotics.

Since the digestive mocus enables the connection between the host and the bacteria that live within it, the investigators would like to characterize the microbiome in the different areas along the digestive system - before antibiotic treatment and after rehabilitation by probiotic treatment versus bacteriotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age: 18 years and up
* Gender: women and men

Exclusion Criteria:

* Pregnancy
* Age under 18 years
* antibiotic treatment 3 months prior to enrollment
* Viral Hepatitis
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-02-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition | 1 year
  stool samples

SECONDARY OUTCOMES:
Microbiome composition | 1 month
  Gastrointestinal tract biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Zamir Halpern, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Department of Gastroentherology, Tel Aviv, Israel